CLINICAL TRIAL: NCT00001941
Title: A Phase I/II Study of the Efficacy and Toxicity of Humanized Anti-Tac (Zenapax(Trademark)) in the Therapy of Tac-Expressing Adult T-Cell Leukemia
Brief Title: Anti-Tac for Treatment of Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Thomas A. Waldmann, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000030; 00-C-0030; NCT00020020 (obsolete NCT alias)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Results first posted 2012-08-09 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: HTLV-I Infection; T Cell Leukemia
Keywords: Interleukin-2 Receptor alpha chain; Interleukin-2; HTLV-I; Adult T-Cell Leukemia (ATL); Monoclonal Antibody (Daclizumab, Zenapax)
MeSH Terms: conditions — HTLV-I Infections; Leukemia, T-Cell; Diabetes Mellitus, Insulin-Dependent, 10; Leukemia-Lymphoma, Adult T-Cell | interventions — Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase I - 2 mg/kg cohort (Experimental): 2 mg/kg daclizumab over 60 minutes intravenously on days 1 and 2
  Interventions: Biological: daclizumab
- Phase I - 4 mg/kg cohort (Experimental): 4 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose
  Interventions: Biological: daclizumab
- Phase I - 6 mg/kg cohort (Experimental): 6 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose
  Interventions: Biological: daclizumab
- Phase I - 8 mg/kg cohort (Experimental): 8 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose
  Interventions: Biological: daclizumab
- Phase II - 8 mg/kg cohort (Experimental): 8 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose
  Interventions: Biological: daclizumab

INTERVENTIONS:
Biological: daclizumab
  Other Names: Zenapax

SUMMARY:
The purpose of the study was to determine: (1) the toxicity and maximum tolerated dose (MTD) of humanized anti-Tac (daclizumab), (Zenapax(Registered Trademark)) in patients with adult T-cell leukemia/lymphoma (ATL); (2) to define the dose of Zenapax(Registered Trademark) required to saturate interleukin 2 receptor alpha (IL-2R) alpha in patients with ATL; (3) determine the clinical response to humanized (Hu) anti-Tac (Zenapax(Registered Trademark) of patients with Tac-expressing adult T-cell leukemia; and (4) determine the serum dieaway curve (pharmacokinetics) of infused humanized (Hu)-anti-Tac in patients who have ATL. This study represented an extension of Metabolism Branch National Cancer Institute (NCI) protocols utilizing modifications of the original murine anti-Tac monoclonal antibody (mAb) developed by our group for the treatment of ATL. The scientific basis for these therapeutic studies is that the leukemic cells of patients with ATL express abnormally high levels of the Tac antigen (IL-2R alpha) on their surface whereas resting normal cells including normal T-cells of the patients do not. One presumed mode of action of Hu-anti-Tac in the treatment of ATL involves the interruption of the interaction of interleukin 2 (IL-2) with its growth factor receptor. To be effective in this goal we must maintain saturation of the IL-2 receptors (IL-2R) with humanized anti-Tac thereby preventing IL-2 mediated proliferation and yielding cytokine deprivation and apoptotic cell death of the leukemic cells. Eligible patients with ATL were treated with escalating doses of Zenapax(Registered Trademark) between groups in the Clinical Center of the National Institutes of Health (NIH). Groups of patients received sufficient Zenapax(Registered Trademark) to yield saturation of the IL-2 receptor for a period of 17 weeks. Clinical response was evaluated using routine immunological and clinical evaluation and by monitoring the saturation of the IL-2R and the absolute number of residual circulating malignant cells by fluorescence activated cell sorting (FACS) analysis using two fluorochrome-labeled non-crossreacting antibodies to the IL-2 receptor, anti-Tac and 7G7/B6, as well as antibodies to cluster of differentiation 3 (CD3), cluster of differentiation 4 (CD4), cluster of differentiation 7 (CD7), and cluster of differentiation 8 (CD8). Furthermore, responses were evaluated in patients with leukemia by Southern blot analysis of the arrangement of the T-cell receptor genes and human T-lymphotropic virus type 1 (HTLV-I) integration. Finally, in select patients, to define the pharmacokinetics of the therapeutic antibody, had planned to monitor the serum levels of the infused Hu-anti-Tac (Zenapax(Registered Trademark)) as a function of time. This study is an essential element of our program involving IL-2R-directed therapeutic studies. If as anticipated the therapy with humanized anti-Tac yields some partial and complete remissions in patients with ATL, we will propose that it be used as a single agent for patients with smoldering and chronic ATL and in association with chemotherapeutic agents to provide a novel approach for the treatment of acute and lymphoma forms of ATL. We also plan a future clinical trial where tentative plans also had been made to evaluate the efficacy and toxicity in ATL patients of saturating doses of Zenapax(Registered Trademark) as compared to identical doses of Zenapax(Registered Trademark) given in association with (90)Y-armed 7G7/B6, a non-competing antibody to IL-2R alpha or in combination with chemotherapy.

DETAILED DESCRIPTION:
Background:

Human T-lymphotropic virus type 1 (HTLV-1)-associated adult T cell leukemia/lymphoma (ATL) is an aggressive lymphoproliferative disorder.

Chemotherapy has had limited impact on survival.

The interleukin 2 receptor alpha (IL-2R alpha) (CD25) is over expressed on ATL cells and the smoldering and chronic stages of ATL are often interleukin 2 (IL-2) dependent.

The monoclonal antibody daclizumab (Zenapax) inhibits interleukin 2 (IL-2) binding to its receptor.

It is hypothesized that daclizumab may inhibit ATL growth.

Objectives:

To determine the toxicity and maximum tolerated dose (MTD) of humanized anti-Tac (daclizumab, Zenapax) in patients with ATL.

To define the dose of Zenapax required to saturate IL-2R alpha in patients with ATL.

To determine the clinical response to humanized (Hu) anti-Tac (Zenapax) of patients with Tac-expressing smoldering and chronic stage adult T cell leukemia.

To determine the serum dieaway curve (pharmacokinetics) of infused humanized (Hu) - anti - Tac in patients who have ATL.

Eligibility:

Smoldering and chronic stage HTLV-1-associated adult T cell leukemia.

At least 5 percent of malignant cells in the peripheral blood or lymph nodes must react with the anti-Tac (CD25) antibody.

Age greater than or equal to 10-years-old.

Patients must have measurable disease.

Patients with and without prior treatment.

Patients must have a granulocyte count of greater than or equal to 500/micro L,

platelets greater than or equal to 25,000/micro L,

and creatinine less than 3.0 gm/dL.

Design:

Phase I patients on cohorts 1-4 received the following: cohort 1: 2 mg/kg over 60 minutes intravenously on days 1 and 2; cohort 2: 4 mg/kg over 90 minutes intravenously on day 1, single dose; cohort 3: 6 mg/kg over 90 minutes intravenously on day 1, single dose; and cohort 4: 8 mg/kg over 90 minutes intravenously on day 1, single dose.

Patients with smoldering or chronic stage ATL will be treated with intravenous daclizumab 8 mg/kg on day 0 and weeks 2, 5, 8, 11 and 14.

Patients achieving a response will continue on treatment with daclizumab 8 mg/kg every 3 weeks for up to 24 months.

Patients achieving a complete response (CR) will continue on treatment with daclizumab 8mg/kg every 3 weeks for up to 24 months.

Patients achieving a partial response (PR) will be maintained on daclizumab 8 mg/kg administered every 3 weeks provided the PR is maintained and no serious adverse event or toxicity related to daclizumab therapy is observed.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Population Base.
* Patients diagnosed with smoldering or chronic human T-lymphotropic virus type 1 (HTLV-I)- associated adult T-cell leukemia.

INCLUSION CRITERIA:

* Patients must have serum antibodies directed to HTLV-I.
* All patients must have a histologically confirmed diagnosis of adult T-cell leukemia/lymphoma.
* At least 5 percent of each patient's peripheral blood, lymph node, pulmonary or dermal malignant cells must react with the anti-Tac mAb as determined by immunofluorescent staining or, alternatively, the serum-soluble interleukin 2 (IL-2) receptor levels must be greater than 1,000 units/ml (normal geometric mean, 235; with a 95% confidence interval of 112 to 502 units/mL).
* Smoldering or chronic stage Tac-expressing adult T-cell leukemia defined by the Shimomyama Criteria (37) are eligible.
* To be diagnosed as smoldering Adult T-cell Leukemia (ATL), the patient must have a normal lymphocyte count (less than 4 times 10^3/mm^3), less than or equal to 5 percent abnormal lymphocytes on morphologic examination of the peripheral blood smear or on fluorescence activated cell sorting (FACS) analysis (cells with a homogenous staining pattern and a greater than 1 log increase in the magnitude of fluorescence emission of the anti-Tac peak over background expression),
* no hypercalcemia,
* lactate dehydrogenase less than or equal to 1.5 times the upper limit of normal,
* no lymphadenopathy,
* no involvement of extra nodal organs except skin or lung and no malignant pleural effusion or ascites.
* If the abnormal lymphocyte count is less than 5 percent, the patient must have at least one histologically proven skin ATL lesion to be diagnosed as smoldering ATL.
* Patients with >5% of circulating lymphocytes that are abnormal are considered to have measurable disease.
* The patient must have a granulocyte count of at least 500/mm^3 and a platelet count of 25,000/mm^3.
* Patients must have a creatinine of less than 3.0 mg/dl.
* Patients must have a Karnofsky performance score of greater than 60 percent.
* ATL patients without, as well as those with, previous chemotherapy will be eligible for inclusion in the study.
* Patients with previous therapy with a monoclonal antibody including anti-Tac will be eligible for the study provided that they do not have a positive HAHA (human antibody to humanized anti-Tac) value (i.e., such patients must have a value greater than 250 ng/ml).
* Omission of cytotoxic chemotherapy for ATL for 3 weeks prior to entry into the trial is required.
* However, patients receiving corticosteroids will not be excluded.
* Patients must have a life expectancy of greater than 2 months.
* Eligible patients must be greater than or equal to 10 years old.
* There is no upper age limit.
* Patients over the age of 18 years must be able to understand and sign an Informed Consent form.
* Eligible minors greater than or equal to 10 years old must give assent to participate in this study.

EXCLUSION CRITERIA:

* Patients with symptomatic central nervous system disease that is due to the adult T-cell leukemia will be excluded.
* However, patients that have both ATL and another HTLV-I-associated disease, tropical spastic paraparesis (TSP), will be included.
* Furthermore, Tac-expressing T cells may be present in the cerebrospinal fluid (CSF) as long as the patient does not have symptomatic central nervous system (CNS) disease.
* Pregnant and/or nursing patients are not eligible for the study.
* Human immunodeficiency virus (HIV) positive patients are excluded from the study.
* Patients with serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) values 5.0-fold greater than the upper limit of normal or bilirubin greater than 2.9 mg/dl will be excluded.
* If a liver function test is judged to be elevated due to the underlying ATL, this parameter will be considered an unevaluable parameter for toxicity determinations.
* Acute or Lymphoma stage HTLV-1 associated adult T cell leukemia.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 1999-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Waldmann, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kohler G, Milstein C. Continuous cultures of fused cells secreting antibody of predefined specificity. Nature. 1975 Aug 7;256(5517):495-7. doi: 10.1038/256495a0. No abstract available. PMID 1172191
- [Background] Levy R, Miller RA. Tumor therapy with monoclonal antibodies. Fed Proc. 1983 Jun;42(9):2650-6. No abstract available. PMID 6343125
- [Background] Catane R, Longo DL. Monoclonal antibodies for cancer therapy. Isr J Med Sci. 1988 Sep-Oct;24(9-10):471-6. PMID 3060441
- [Background] Hakimi J, Chizzonite R, Luke DR, Familletti PC, Bailon P, Kondas JA, Pilson RS, Lin P, Weber DV, Spence C, et al. Reduced immunogenicity and improved pharmacokinetics of humanized anti-Tac in cynomolgus monkeys. J Immunol. 1991 Aug 15;147(4):1352-9. PMID 1869828
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-C-0030.html
- See also: World Health Organization (WHO) — http://whqlibdoc.who.int/offset/WHO_OFFSET_48.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase II- 8 mg/kg Cohort: 8 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose
Period: Overall Study
Arm/Group | Phase I - 2 mg/kg Cohort | Phase I - 4 mg/kg Cohort | Phase I - 6 mg/kg Cohort | Phase I - 8 mg/kg Cohort | Phase II- 8 mg/kg Cohort
Started | 3 | 5 | 3 | 3 | 20
Completed | 3 | 5 | 3 | 3 | 19
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — not treated- rapidly progressing disease | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I & II Cohorts (2-8 mg/kg): Phase I - 2 mg/kg cohort 2 mg/kg daclizumab over 60 minutes intravenously on days 1 and 2 Phase I - 4 mg/kg cohort 4 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose Phase I - 6 mg/kg cohort 6 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose Phase I - 8 mg/kg cohort 8 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose Phase II- 8 mg/kg cohort 8 mg/kg daclizumab over 90 minutes intravenously on day 1, single dose
Arm/Group | Phase I & II Cohorts (2-8 mg/kg)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 29
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 47.37 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 25
  Hispanic | 2
  White | 6
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Duration of Response
Description: Duration of response was defined as the interval from the time response is first achieved to the time progression from the best response is detected. Responses are assessed by a modified World Health Organization (WHO) criteria. Partial response is a reduction of >=50% saturation in the circulating leukemic cell count; complete response is disappearance of all measurable and non-measurable disease lasting more than 1 month; stable disease is patients who did not meet the criteria; and progressive disease is a >=25% increase in leukemic cell count.
Time Frame: 21-220 weeks
Population: Phase I is not reported because phase I studies only determine maximum tolerated dose.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Phase II- 8 mg/kg Cohort
Number analyzed (Participants) | 19
Weeks | 114 [21 to 220]

2. Primary Outcome: Overall Survival
Description: Measured from the time the patient is consented until death.
Time Frame: 132.6 weeks
Population: Phase I is not reported because phase I studies only determine maximum tolerated dose.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Phase II- 8 mg/kg Cohort
Number analyzed (Participants) | 19
Weeks | 132.6 [53.9 to NA] — The upper end of the confidence interval was not reached because at last follow-up a patient had an ongoing response at last contact.

3. Primary Outcome: Percentage of Participants With an Overall Response Rate
Description: Participants overall response rate was defined as complete response (CR) + partial response (PR) from study consent until progression was measured. Responses was assessed by a modified World Health Organization (WHO) criteria. Partial response is a reduction of >=50% saturation in the circulating leukemic cell count; complete response is disappearance of all measurable and non-measurable disease lasting more than 1 month; and progressive disease is a >=25% increase in leukemic cell count
Time Frame: up to 220 weeks
Population: Phase I is not reported because phase I studies only determine maximum tolerated dose.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase II- 8 mg/kg Cohort
Number analyzed (Participants) | 19
Percentage of participants | 20

4. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 12 months
Population: Data is not available separately per cohort.
Measure: Number; unit: Participants
Arm/Group | Phase I & II Cohorts (2-8 mg/kg)
Number analyzed (Participants) | 34
Participants | 32

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Phase II- 8 mg/kg Cohort
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II- 8 mg/kg Cohort (N=34)
Cardiovascular/Arrhythmia -Other (Specify, congestive heart failure (CHF)) (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II- 8 mg/kg Cohort (N=34)
Amylase (Investigations) | 4 (25)
CPK (creatine phosphokinase) (Investigations) | 1 (1)
Leukocytes (total white blood count (WBC)) (Investigations) | 4 (24)
Lymphopenia (Investigations) | 3 (13)
Neutrophils/granulocytes (absolute neutrophil count (ANC)/absolute granulocyte count (AGC)) (Investigations) | 4 (22)
Partial thromboplastin time (PTT) (Investigations) | 1 (1)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 2 (2)
Edema (General disorders) | 1 (1) — feet edema mild edema in lower extremities edema legs
Flatulence (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Investigations) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypercholesterolemia (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (13)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3)
Dermatology/Skin-Other (Specify, Lesions Lt elbow) (Skin and subcutaneous tissue disorders) | 1 (1)
Lipase (Investigations) | 2 (2)
Wound-non-infectious (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 1 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (4)
Prothrombin time (PT) (Investigations) | 2 (12)
Headache (Nervous system disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 3 (3)
Pulmonary-Other (Specify, URI (upper respiratory infection)) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal/Genitourinary-Other (Specify, UTI (urinary tract infection)) (Renal and urinary disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Neuropathy-sensory (Nervous system disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 2 (2)
Bilirubin (Hepatobiliary disorders) | 2 (7)
Creatinine (Investigations) | 2 (3)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 2 (3)
Dyspepsia/heartburn (Gastrointestinal disorders) | 1 (1)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (2)
Earache (otalgia) (Ear and labyrinth disorders) | 1 (1)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (3)
SGOT (aspartate aminotransferase (AST)) (serum glutamic oxaloacetic transaminase) (Investigations) | 6 (8)
SGPT (alanine aminotransferase (ALT)) (serum glutamic pyruvic transaminase) (Investigations) | 5 (7)
Vomiting (Gastrointestinal disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (8)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (2)
Pain-Other (Specify, sore throat pain ; rt knee pain) (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was closed to accrual since the cessation of the production of daclizumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No